CLINICAL TRIAL: NCT01627886
Title: Open-Label, Balanced, Randomized,Two-Treatment, Two-Sequence, Two-Period, Single-Dose, Crossover Oral Bioequivalence Study Of Ibandronate Sodium 150 mg Tablets Of Dr. Reddy's Laboratories Limited, India and 'BONIVA®' 150 mg (Ibandronate Sodium) Tablets Of Roche Laboratories Inc., USA In Healthy, Adult, Human Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Ibandronate Sodium Tablets 150 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BA0859144-01
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2008-11

CONDITIONS: Healthy
Keywords: Bioequivalence; Ibandronate Sodium; crossover
MeSH Terms: interventions — Ibandronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibandronate sodium tablets 150 mg (Experimental): Ibandronate sodium tablets 150 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Ibandronate sodium
- Boniva (Active Comparator): Boniva Tablets 150 mg of Roche Laboratories Inc, USA
  Interventions: Drug: Ibandronate sodium

INTERVENTIONS:
Drug: Ibandronate sodium — Ibandronate sodium Tablets 150 mg
  Other Names: Boniva

SUMMARY:
This is an open label, randomised, balanced, two-treatment, two-period, two-sequence, crossover, oral bioequivalence study.

DETAILED DESCRIPTION:
Open-Label, Balanced, Randomized,Two-Treatment, Two-Sequence, Two-Period, Single-Dose, Crossover Oral Bioequivalence Study Of Ibandronate Sodium 150 mg Tablets Of Dr. Reddy's Laboratories Limited, India And 'BONIVA®' 150 mg (Ibandronate Sodium)Tablets Of Roche Laboratories Inc., USA In Healthy, Adult, Human Subjects Under Fasting Conditions (With As Many Postmenopausal Women As Possible).

ELIGIBILITY:
Inclusion Criteria:

1. The subjects should be healthy human of 18 years or older.
2. The subjects should be screened within 21 days prior to the administration of first dose of the study drug.
3. The subjects should have a BMI between 19 and 30 weight in kg/ height2 in meter.
4. The subjects should be able to communicate effectively with study personnel.
5. The subjects should be able to give written informed consent to participate in the study.

   If subject is a female volunteer and
6. Is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms,foams, jellies, diaphragm, intrauterine device (IUD), or abstinence or
7. Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject) or
8. Should be postmenopausal healthy women who have attained complete menopause and have not had menstruation for at least one year and are not on hormone replacement therapy.
9. Should have 17ß-estradiol serum levels of ≤92 pmol/L, follicle stimulating hormone (FSH) of ≥40 IU/L during the screening (only for postmenopausal healthy women)

Exclusion Criteria:

1. The subjects who have a history of allergic responses to Ibandronate or other related drugs.
2. The subjects who have significant diseases or clinically significant abnormal findings during screening [medical history, physical examination, laboratory evaluations, ECG, X-ray and vaginal ultrasonography recordings (only for female subjects)]
3. The subjects who have any disease or condition which might compromise the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system, diabetes, psychosis or any other body system.
4. The subjects who have a history or presence of bronchial asthma.
5. The subject who have used enzyme-modifying drugs within 30 days prior to receiving the first dose of study medication.
6. The subjects who have history of drug dependence, recent history of alcoholism or of moderate alcohol uses.
7. The subjects who are smokers who smoke more than or equal to 10 cigarettes per day or more than or equal to 20 biddies per day or those who can not refrain from smoking during study period.
8. The subjects with a history of difficulty with donating blood or difficulty in accessibility of veins.
9. The subjects who have donated 1 unit (350 ml / 450 ml) blood within 90 days prior to receiving the first dose of study medication.
10. The subjects who have a positive hepatitis screen (includes subtypes A, B, C & E).
11. The subjects who have a positive test result for HIV antibody and / or syphilis (RPR/VDRL).
12. The subject who receives an investigational product, or has participated in a drug research study within a period of 90 days prior to the first dose of the study medication administration.
13. Female volunteers demonstrating a positive pregnancy screen.
14. Female volunteers who are currently breast-feeding.
15. Female volunteers not willing to use contraception during the study.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2008-09; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Area under curve(AUC) | Prior to dosing (0.0 hour) and at 0.25, 0.50, 0.75, 1.0, 1.25, 1.50, 2.0, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 10.0, 12.0, 24.0, 36.0, 48.0 and 72.0 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Simran Sethi, MBBS, Principal Investigator — BA Research India Ltd
Locations (1):
- BA Research India Ltd, Ahmedabad, Gujarat, India